CLINICAL TRIAL: NCT01710579
Title: Ano-rectal 3D High Resolution Manometry: Normal Values and Comparison With Ultrasound Examination in Healthy Volunteers, Patients With Fecal Incontinence and Patients With Constipation
Brief Title: Normal Values in Ano-rectal 3D High Resolution Manometry
Acronym: NOMAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.729
Record Dates: First submitted 2012-09-14; First posted 2012-10-19 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2012-09

CONDITIONS: Anorectal Disorder; Fecal Incontinence; Constipation
Keywords: Primary esophageal achalasia; endoscopic myotomy; high resolution manometry
MeSH Terms: conditions — Rectal Diseases; Fecal Incontinence; Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ARM 1 Healthy Volunteers (Other): Ano-rectal 3D high resolution manometry, ano-rectal radial endsonography, dynamic ano-rectal endosonography
  Interventions: Procedure: Anorectal 3D-high resolution manometry; Procedure: Anorectal radial endosonography (rotative 360° probe); Procedure: Dynamic anorectal endosonography (sagittal and radial)
- ARM 2: Patients with fecal incontinence (Other): Ano-rectal 3D high resolution manometry, ano-rectal radial endsonography, dynamic ano-rectal endosonography
  Interventions: Procedure: Anorectal 3D-high resolution manometry; Procedure: Anorectal radial endosonography (rotative 360° probe); Procedure: Dynamic anorectal endosonography (sagittal and radial)
- ARM 3 Patients with constipation (Other): Ano-rectal 3D high resolution manometry, ano-rectal radial endsonography, dynamic ano-rectal endosonography
  Interventions: Procedure: Anorectal 3D-high resolution manometry; Procedure: Anorectal radial endosonography (rotative 360° probe); Procedure: Dynamic anorectal endosonography (sagittal and radial)

INTERVENTIONS:
Procedure: Anorectal 3D-high resolution manometry — Anorectal probe is used with a single-use protective sheath with an inflation balloon Control of balloon deflation Patient in left lateral decubitus position with hips flexed to 90° (this position is the most commonly use and the most convenient) Transanal insertion 2 minutes resting period: resting anal pressure will be evaluated the second minute of rest Sustained voluntary maximal squeeze for at least 30 seconds; the maneuver will be repeated once Valsalva Bear down maneuver; the maneuver will be repeated once Anorectal reflexes evaluation with 20-, 40- and 60-ml intra-rectal balloon inflation Probe removal
Procedure: Anorectal radial endosonography (rotative 360° probe) — Patient in left lateral decubitus position with hips flexed to 90° Transanal probe insertion Evaluation of internal and external anal sphincter integrity and puborectalis muscle at rest
Procedure: Dynamic anorectal endosonography (sagittal and radial) — Patient in left lateral decubitus position with hips flexed to 90° Rectum is filled with 50-ml water Probe is covered with a water-filled balloon to maintain the acoustic window for the ultrasound wave Transanal probe insertion Slow and manual rotation of the linear probe through 360° to identify the various layers constituting the anal wall (mucosa, IAS, EAS), the layer forming the rectal wall and the perirectal tissues (puborectalis muscle, bladder, and vagina or prostate) After the initial examination, the patient will be asked to make a defecation effort with the probe left in the same position

SUMMARY:
Ano-rectal manometry is indicative in patients with either fecal incontinence or constipation. Recently anorectal 3D- high resolution manometry has been developed. Pressure variations are measured circumferentially along the anal canal. It may allow a better understanding of anorectal disorders by displaying anal pressure asymmetry and it could be useful to assess the functional anatomy of the pelvic floor better than conventional manometry.

ELIGIBILITY:
Arm 1: 50 healthy volunteers Inclusions will be stratified on gender (10 males, 40 females), age (15 subjects under 40 years; 20 subjects between 40 and 60 years; and 15 subjects >60 years) and parous (10 nullipara and 30 parous women).

Inclusion criteria:

Subject older than 18 years Absence of anorectal symptoms (no constipation, no fecal incontinence) Absence of pelvic floor disorders Vaizey score = 0 Kess score < 9 Subject with health insurance Written informed consent Non inclusion criteria: Patient younger than 18 years Pregnancy Incapability to give consent No written informed consent Participation to another study at the same time Previous ano-rectal surgery Pelvic radiotherapy Neurological disorder Diabetes mellitus

Arm 2: 50 patients with fecal incontinence

Inclusion criteria:

Subject older than 18 years Patient referred for anorectal manometry and/or ultrasound examination Fecal incontinence as main complain Vaizey score > 6 Kess score < 9 Subject with health insurance Written informed consent

Non inclusion criteria:

Patient younger than 18 years Pregnancy Incapability to give consent No written informed consent Participation to another study at the same time Rectal tumor Rectal stenosis Ileo-anal or ileo-rectal anastomosis Anal fissure Anal fistula Arm 3: 50 patients with constipation

Inclusion criteria:

Subject older than 18 years Patient referred for anorectal manometry and/or ultrasound examination Constipation as main complain Feeling of incomplete evacuation and/or manual disimpaction defined as needing to press in or around the anus to aid defecation Vaizey score < 6 Kess score < 9 Subject with health insurance Written informed consent

Non inclusion criteria:

Patient younger than 18 years Pregnancy Incapability to give consent No written informed consent Participation to another study at the same time Rectal tumor Rectal stenosis Ileo-anal or ileo-rectal anastomosis Anal fissure Anal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Anal pressure pattern at rest, during voluntary maximal squeezing and bear down Anal pressure pattern at rest, during voluntary maximal squeezing and bear down | during procedure
  Following parameters will be measured at the level of anal sphincter:
  * Minimal pressure (amplitude and location)
  * Maximal pressure (amplitude and location)
  * Mean pressure
  * Asymmetry

SECONDARY OUTCOMES:
presence of ano-rectal reflex. | during procedure
Ano-rectal radial endosonography | During procedure
  Evaluation of internal and external anal sphincter integrity and puborectalis muscle at rest
Dynamic ano-rectal endoconography | During procedure
  presence of pelvic floor disorder (rectocele, enterocele)

CONTACTS AND LOCATIONS:
Locations (1):
- Unité d'Exploration Fonctionnelle Digestive Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Result] Mion F, Garros A, Brochard C, Vitton V, Ropert A, Bouvier M, Damon H, Siproudhis L, Roman S. 3D High-definition anorectal manometry: Values obtained in asymptomatic volunteers, fecal incontinence and chronic constipation. Results of a prospective multicenter study (NOMAD). Neurogastroenterol Motil. 2017 Aug;29(8). doi: 10.1111/nmo.13049. Epub 2017 Mar 2. PMID 28251732